CLINICAL TRIAL: NCT05121467
Title: Muscular Endurance And Its Association With Neck Pain, Disability, Neck Awareness, And Kinesiophobia In Patients With Cervical Disc Herniation
Brief Title: Muscular Endurance And Its Association With Neck Pain, Disability, Neck Awareness, And Kinesiophobia
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Tuğba DERE, Physiotherapist, Hacettepe University
Other Study IDs: 200415001
Record Dates: First submitted 2021-05-27; First posted 2021-11-16 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Cervical Disc Herniation
Keywords: Degenerative Disc Disease; Cervical Spine; Neck Pain; Muscles
MeSH Terms: conditions — Intervertebral Disc Degeneration; Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Cervical Disc Herniation: Endurance tests were performed for 9 muscles/muscle groups in the cervical and scapular regions, upper limb, and trunk Visual Analogue Scale (VAS) and Neck Disability Index (NDI) Fremantle Neck Awareness Questionnaire (FreNAQ) Tampa Scale of Kinesiophobia (TSK)
  Interventions: Other: Pain Assessment; Other: Assessment of Muscular Endurance; Other: Assessment of Neck Awareness; Other: Assessment of Fear of Movement

INTERVENTIONS:
Other: Pain Assessment — Visual Analogue Scale (VAS) were included in the study
Other: Assessment of Muscular Endurance — The endurance of the 9 muscles/muscle groups including cervical flexor, extensor, deep flexor muscles, trunk flexor, extensor, lateral flexor, and stabilizer muscles, upper extremity, and scapular muscles (mm. serratus anterior and trapezius) were evaluated based on the assessment instructions given in the studies of Edmonston et al., Grimmer et al., Evans et al., Reece et al., ACSM guideline
Other: Assessment of Neck Awareness — The Turkish version of the Fremantle Neck Awareness Questionnaire (FreNAQ) which was developed by Wand et al. to assess neck awareness in patients with chronic neck pain was used in this study
Other: Assessment of Fear of Movement — The fear of movement was assessed by the Turkish version of the Tampa Scale of Kinesiophobia which originally developed by Kori et al.

SUMMARY:
The aim of this study was to investigate the relationship of muscular endurance of the trunk, upper extremities, and scapular region as well as cervical region, with pain, neck awareness, and kinesiophobia in patients with cervical disc herniation. Thirty-six patients between 18-65 years with a diagnosis of cervical disc herniation and having neck pain of 2 and above at rest according to the Visual Analogue Scale (VAS) were included in the study. After the evaluation of musculoskeletal system, endurance tests were performed for 9 muscles/muscle groups in the cervical and scapular regions, upper limb, and trunk. Pain severity was measured by VAS and Neck Disability Index (NDI), neck awareness with Fremantle Neck Awareness Questionnaire (FreNAQ), and fear of movement with Tampa Kinesiophobia Scale (TKS).

DETAILED DESCRIPTION:
Cervical disc herniation occurs as a result of a sudden trauma or chemical/mechanical degenerative changes in the cervical spine, and is more common in women. The most common age range for disc herniation is 51-60 years with the increase in prevalence with age in both genders, and the most affected disc level is C6-C7. The clinical presentation such as weakness in cervical musculature, decreased endurance, loss of motor control and postural stabilization, changes in reflexes, loss of sensation, and movement limitations varies based on the location of the disc. The pain caused by any damage or compression in the cervical spinal nerve root is seen along the affected nerve dermatome as well as the head, neck, scapula, shoulder, and upper extremity, and accompanied by spasm in the cervical muscles.

Cervical muscles have a large number of sensory receptors responsible for vestibular, visual, and postural control by the deep suboccipital muscles with dense muscle spindles. They are responsible for the stabilization of the head, neck, and the thoracic region against involuntary perturbation by maintaining the continuity of the posture; they ensure the mobility of neck and upper limbs, and contribute neck awareness and postural reflexes. Intense proprioceptive receptors of deep cervical muscles support the motor control of the trunk muscles, mutually trunk muscles contribute to stabilization of the head and neck; and through the thoracolumbar fascia they work in coordination with scapular muscles. It has been known that any involvement of cervical, trunk, and scapular region muscles, as a whole, contribute to the etiology of the neck pain in patients due to their strong anatomical relations. In addition, the contribution of the upper extremity muscles in the stabilization of the cervical spine and the triggering of neck pain during upper extremity movements also reveal the importance of the motor control of upper extremity muscles in these patients.

Endurance of the cervical muscles has been known to have more responsibility on the spinal stabilization than strength in patients with chronic neck pain, causing an increase in pain with the decrease in endurance. In cervical disc herniation, the pathology in the cervical region causing the malalignment of the spine not only deteriorate the strength and endurance of the neck muscles, but it also affects other muscles around the spine. Further, proprioceptive receptors in the cervical muscles lose the ability to detect changes in muscle tension due to the reduced endurance, which in turn affect neck awareness. On the other hand, since chronic pain is closely related to cognitive and behavioral factors, pain worsens as a result of activity avoidance according to the fear-avoidance model, hence the kinesiophobia also increases by the decrease in cervical muscle endurance in chronic neck pain.

Recent studies revealed the connection between the endurance of neck muscles and pain, neck awareness, and fear of movement in patients with cervical disc herniation in literature. However, the evidence related to the relation between scapular, upper extremities, and trunk muscles' endurance and neck pain, neck awareness, and fear of movement has still been lacking. Therefore, the aim of the present study was to investigate the association between the endurance of these muscles and neck pain, neck awareness, and kinesiophobia in patients with cervical disc herniation.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of cervical disc herniation confirmed by MR radiography, direct radiography, and clinical and physical examination
2. Having neck pain at rest for 3 months or more with a severity of 2 or above according to the Visual Analogue Scale (VAS)
3. Having a score of 5 or more from the NDI
4. Being able to comply with the instructions of the physiotherapist

Exclusion Criteria:

1. Patients with spinal tumors/deformities/congenital malformations
2. Who underwent cervical or upper extremity surgery in the previous 6 months were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was carried out by patients who were diagnosed with cervical disc herniation and directed to Hacettepe University, Faculty of Physical Medicine and Rehabilitation for physical therapy consultation. The patients who met the inclusion criteria were given detailed information about the study, and signed a consent form.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Neck Flexor Muscular Endurance | two weeks
  The endurance of the neck flexor muscles was evaluated by elevating the head of the patient 6 cm in the supine hook position. With the removal of the head support, the maximum time spent in this position was recorded in seconds. The test was ceased when a 5-degree deviation seen in the goniometer which followed the vertical angle of the mandible.
Assessment of Neck Extensor Muscular Endurance | two weeks
  Neck extensor muscle endurance was evaluated in prone position hanging the head and neck from the bed and placing the arms of the patients on side of the body. A 2 kg-weight (sandbag) was placed behind the head with a Velcro corresponding to the C6 level. The maximum time spent holding the head in neutral position was recorded in seconds.
Assessment of Cervical Deep Flexor Muscular Endurance | two weeks
  Cervical deep flexor muscle endurance was evaluated in the supine hook position by asking the patients to put their hands on their abdomen, look at the chest level by pulling their chin inward and raising their head 2.5 cm from the bed. The maximum time spent to hold their head in this position was recorded.
Assessment of Trunk Flexor Muscular Endurance | two weeks
  In order to evaluate the trunk flexor muscle endurance, the patients were asked to hold their hands on the opposite shoulders in the supine hook position. Then, they were asked to lift up the upper body until the lower end of the scapula lifted off the ground, and the maximum time spent to keep the position was recorded in seconds.
Assessment of Trunk Extensor Muscular Endurance | two weeks
  Endurance of the trunk extensor muscles was evaluated in prone position hanging the upper body from the bed from the level of spina iliaca anterior superior. The lower limb was fixed by the evaluator. The participants were asked to bring both hands together on their neck and lift their body parallel to the ground. The maximum time spent to hold the position was noted in seconds.
Assessment of Trunk Lateral Flexor Muscular Endurance | two weeks
  Endurance of the trunk lateral flexor muscles was assessed in a side-lying position and participants were asked to pull their knees gently on their abdomen. The upper leg was placed in front of the other foot. The body weight was carried on the forearm and feet, and the upper hand was placed on the opposite shoulder. Then, the patients were asked to elevate the hip until the pelvis and trunk reached a horizontal position. Measurements were made for each side, and the maximum time spent to maintain the position was recorded in seconds.
Assessment of Trunk Stabilizer Muscular Endurance | two weeks
  The endurance of the trunk stabilizer muscles was evaluated in prone by the bridge test. The patients were initially asked to place in the prone position supported on the knee and forearms. Then, they were asked to stand on their forearms and toes by raising their knees and maintain this position. The time they held the position was noted in seconds.
Assessment of Upper Extremity Muscular Endurance | two weeks
  Upper extremity muscular endurance was evaluated in a modified push-ups exercise position. Hands were placed shoulder-width apart on the ground, and the trunk was asked to be closer to the ground with elbow flexion in the prone position. Care was given to hold the body weight on the knees and hands. The number of repetitions for 30 seconds was noted.
Assessment of M. serratus anterior and m. trapezius Muscular Endurance | two weeks
  M. serratus anterior and m. trapezius muscles' endurance were evaluated via the scapular muscle endurance test. The patient was placed in standing position with shoulder and elbow flexed at 90°. A dynamometer (Feta 0202 1kg/10N) with a resistance of 1kg/10N was placed between hands by placing a 30 cm ruler between the elbows. The patients were asked to hold the dynamometer in the position that they would be most comfortable, and bring their shoulders to external rotation, and pull it with both hands. The time in which they were able to hold the position without dropping the ruler was noted in seconds.
Assessment of Level of Pain | two weeks
  In order to evaluate the pain levels of the patients, Visual Analogue Scale (VAS), which was developed by Price et al. to evaluate the pain level of patients with chronic pain, was used.19 Patients were asked to rate their neck pain on the 10 cm horizontal line where "0" meant no pain, and "10" meant the most severe pain. The points that patients marked were measured with a ruler and noted as pain severity at resting, during activity, and night, separately.
Assessment of Neck Awareness | two weeks
  The Turkish version of the Fremantle Neck Awareness Questionnaire (FreNAQ) which was developed by Wand et al. to assess neck awareness in patients with chronic neck pain was used in this study. The FreNAQ consists of 9 items related to neck pain, attention, and proprioceptive awareness. Each question is scored between 0 and 4 (0 = Never / I never feel this way, 1 = I rarely feel this way, 2 = I sometimes feel this way, 3 = I often feel this way, 4 = I often or always feel this way). The total score of the questionnaire is between 0 and 36. Higher scores indicate higher degrees of neck awareness
Assessment of Fear of Movement | two weeks
  The fear of movement was assessed by the Turkish version of the Tampa Scale of Kinesiophobia which originally developed by Kori et al. The questionnaire which evaluates injury avoidance and fear of movement consists of 17 items, and each item is scored between 1 and 4 (1 = Strongly disagree, 4 = Strongly agree). The total score ranges from 17 to 68. Higher scores indicate a higher kinesiophobia level.
Assessment of Disability | two weeks
  The NDI was developed as the neck version of the Oswestry Low Back Pain Disability Questionnaire to evaluate the disability caused by chronic neck pain. Each question is scored between 0 and 5 and the level of disability of the patients is classified according to the following scoring; 0-4 points, no disability; 5-14 points, mild disability; 14-24 points, moderate disability; 25-34 points, severe disability; and, 35-50 points, complete disability.

CONTACTS AND LOCATIONS:
Overall Officials: İpek A GÜRBÜZ, Ass. Prof., Principal Investigator
Locations (1):
- Tuğba, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hammer C, Heller J, Kepler C, editors. Epidemiology and pathophysiology of cervical disc herniation. Seminars in Spine Surgery; 2016: Elsevier.
- [Background] Kumagai G, Wada K, Kudo H, Asari T, Chiba D, Ota S, Takeda O, Koyama K, Nakaji S, Ishibashi Y. Associations between cervical disc degeneration and muscle strength in a cross-sectional population-based study. PLoS One. 2019 Jan 25;14(1):e0210802. doi: 10.1371/journal.pone.0210802. eCollection 2019. PMID 30682082
- [Background] Sharrak S, Al Khalili YJS. Cervical disc herniation. 2020.
- [Background] Carette S, Fehlings MG. Clinical practice. Cervical radiculopathy. N Engl J Med. 2005 Jul 28;353(4):392-9. doi: 10.1056/NEJMcp043887. No abstract available. PMID 16049211
- [Background] Zabihhosseinian M, Holmes MW, Murphy B. Neck muscle fatigue alters upper limb proprioception. Exp Brain Res. 2015 May;233(5):1663-75. doi: 10.1007/s00221-015-4240-x. Epub 2015 Mar 13. PMID 25764200
- [Background] Kim JB, Yun CK, Lee MH. A comparison of the shoulder and trunk muscle activity according to the various resistance condition during push up plus in four point kneeling. J Phys Ther Sci. 2017 Jan;29(1):35-37. doi: 10.1589/jpts.29.35. Epub 2017 Jan 30. PMID 28210034
- [Background] Cromwell RL, Aadland-Monahan TK, Nelson AT, Stern-Sylvestre SM, Seder B. Sagittal plane analysis of head, neck, and trunk kinematics and electromyographic activity during locomotion. J Orthop Sports Phys Ther. 2001 May;31(5):255-62. doi: 10.2519/jospt.2001.31.5.255. PMID 11352192
- [Background] Gong W, Kim C, Lee YJJoPTS. Correlations between cervical lordosis, forward head posture, cervical ROM and the strength and endurance of the deep neck flexor muscles in college students. 2012;24(3):275-7.
- [Background] Darnell MW. A proposed chronology of events for forward head posture. J Craniomandibular Pract. 1983 Sep-Nov;1(4):49-54. doi: 10.1080/07345410.1983.11677844. No abstract available. PMID 6586880
- [Background] Vaegter HB, Madsen AB, Handberg G, Graven-Nielsen T. Kinesiophobia is associated with pain intensity but not pain sensitivity before and after exercise: an explorative analysis. Physiotherapy. 2018 Jun;104(2):187-193. doi: 10.1016/j.physio.2017.10.001. Epub 2017 Oct 28. PMID 29290378
- [Background] Boersma K, Linton SJ. Psychological processes underlying the development of a chronic pain problem: a prospective study of the relationship between profiles of psychological variables in the fear-avoidance model and disability. Clin J Pain. 2006 Feb;22(2):160-6. doi: 10.1097/01.ajp.0000159582.37750.39. PMID 16428950
- [Background] Woodhouse A, Vasseljen O. Altered motor control patterns in whiplash and chronic neck pain. BMC Musculoskelet Disord. 2008 Jun 20;9:90. doi: 10.1186/1471-2474-9-90. PMID 18570647
- [Background] Falla DL. Neuromuscular control of the cervical spine in neck pain disorders. Fundamentals of Musculoskeletal Pain: IASP Press; 2008. p. 417-30.
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Aslan E, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagly N. The cultural adaptation, reliability and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2008 May 15;33(11):E362-5. doi: 10.1097/BRS.0b013e31817144e1. PMID 18469684
- [Background] Neumanm DA. Kinesiology of the musculoskeletal system: foundations for physical rehabilitation: Mosby; 2002.
- [Background] Edmondston SJ, Wallumrod ME, Macleid F, Kvamme LS, Joebges S, Brabham GC. Reliability of isometric muscle endurance tests in subjects with postural neck pain. J Manipulative Physiol Ther. 2008 Jun;31(5):348-54. doi: 10.1016/j.jmpt.2008.04.010. PMID 18558277
- [Background] Grimmer K. Measuring the endurance capacity of the cervical short flexor muscle group. Aust J Physiother. 1994;40(4):251-4. doi: 10.1016/S0004-9514(14)60461-X. PMID 25025606
- [Background] Evans K, Refshauge KM, Adams R. Trunk muscle endurance tests: reliability, and gender differences in athletes. J Sci Med Sport. 2007 Dec;10(6):447-55. doi: 10.1016/j.jsams.2006.09.003. Epub 2006 Dec 1. PMID 17141568
- [Background] Reece JD. Development of a prone bridge test as a measurement of abdominal stability in healthy adults. 2009.
- [Background] Negrete RJ, Hanney WJ, Kolber MJ, Davies GJ, Ansley MK, McBride AB, Overstreet AL. Reliability, minimal detectable change, and normative values for tests of upper extremity function and power. J Strength Cond Res. 2010 Dec;24(12):3318-25. doi: 10.1519/JSC.0b013e3181e7259c. PMID 21088548
- [Background] ONAN D. Kronik Boyun Ağrılı Hastalarda Boyun Farkındalığının, Fremantle Boyun Farkındalık Anketi İle Değerlendirilmesi: Türkçe Versiyon, Geçerlilik ve Güvenirlik Çalışması. 2018.
- [Background] Wand BM, Catley MJ, Rabey MI, O'Sullivan PB, O'Connell NE, Smith AJ. Disrupted Self-Perception in People With Chronic Low Back Pain. Further Evaluation of the Fremantle Back Awareness Questionnaire. J Pain. 2016 Sep;17(9):1001-12. doi: 10.1016/j.jpain.2016.06.003. Epub 2016 Jun 18. PMID 27327235
- [Background] Yilmaz ÖT, Yakut Y, Uygur F, Uluğ NJFR. Tampa Kinezyofobi Ölçeği'nin Türkçe versiyonu ve test-tekrar test güvenirliği. 2011;22(1):44-9.
- [Background] Overholser BR, Sowinski KM. Biostatistics primer: part 2. Nutr Clin Pract. 2008 Feb;23(1):76-84. doi: 10.1177/011542650802300176. PMID 18203967
- [Background] James WP. WHO recognition of the global obesity epidemic. Int J Obes (Lond). 2008 Dec;32 Suppl 7:S120-6. doi: 10.1038/ijo.2008.247. PMID 19136980
- [Background] Arslan T. Müzisyenlerde üst ekstremite fonksiyonlarının değerlendirilmesi: Eastern Mediterranean University EMU; 2017.
- [Background] Ghamkhar L, Kahlaee AH. The effect of trunk muscle fatigue on postural control of upright stance: A systematic review. Gait Posture. 2019 Jul;72:167-174. doi: 10.1016/j.gaitpost.2019.06.010. Epub 2019 Jun 11. PMID 31207565
- [Background] Im B, Kim Y, Chung Y, Hwang S. Effects of scapular stabilization exercise on neck posture and muscle activation in individuals with neck pain and forward head posture. J Phys Ther Sci. 2016 Mar;28(3):951-5. doi: 10.1589/jpts.28.951. Epub 2016 Mar 31. PMID 27134391
- [Background] Falla D, Bilenkij G, Jull G. Patients with chronic neck pain demonstrate altered patterns of muscle activation during performance of a functional upper limb task. Spine (Phila Pa 1976). 2004 Jul 1;29(13):1436-40. doi: 10.1097/01.brs.0000128759.02487.bf. PMID 15223935
- [Background] Lin JJ, Lim HK, Soto-quijano DA, Hanten WP, Olson SL, Roddey TS, Sherwood AM. Altered patterns of muscle activation during performance of four functional tasks in patients with shoulder disorders: interpretation from voluntary response index. J Electromyogr Kinesiol. 2006 Oct;16(5):458-68. doi: 10.1016/j.jelekin.2005.09.008. Epub 2005 Dec 1. PMID 16324850
- [Background] Hlavenka TM, Christner VFK, Gregory DE. Neck posture during lifting and its effect on trunk muscle activation and lumbar spine posture. Appl Ergon. 2017 Jul;62:28-33. doi: 10.1016/j.apergo.2017.02.006. Epub 2017 Feb 27. PMID 28411737
- [Background] Falla D, Farina D. Neural and muscular factors associated with motor impairment in neck pain. Curr Rheumatol Rep. 2007 Dec;9(6):497-502. doi: 10.1007/s11926-007-0080-4. PMID 18177604
- [Background] Lee H, Nicholson LL, Adams RD. Neck muscle endurance, self-report, and range of motion data from subjects with treated and untreated neck pain. J Manipulative Physiol Ther. 2005 Jan;28(1):25-32. doi: 10.1016/j.jmpt.2004.12.005. PMID 15726032
- [Background] Ariens GA, Bongers PM, Douwes M, Miedema MC, Hoogendoorn WE, van der Wal G, Bouter LM, van Mechelen W. Are neck flexion, neck rotation, and sitting at work risk factors for neck pain? Results of a prospective cohort study. Occup Environ Med. 2001 Mar;58(3):200-7. doi: 10.1136/oem.58.3.200. PMID 11171934
- [Background] Jull G, Falla D, Treleaven J, Sterling M, O'Leary S. A therapeutic exercise approach for cervical disorders. 2004
- [Background] Castelein B, Cools A, Bostyn E, Delemarre J, Lemahieu T, Cagnie B. Analysis of scapular muscle EMG activity in patients with idiopathic neck pain: a systematic review. J Electromyogr Kinesiol. 2015 Apr;25(2):371-86. doi: 10.1016/j.jelekin.2015.01.006. Epub 2015 Jan 31. PMID 25683111
- [Background] Peolsson A, Kjellman G. Neck muscle endurance in nonspecific patients with neck pain and in patients after anterior cervical decompression and fusion. J Manipulative Physiol Ther. 2007 Jun;30(5):343-50. doi: 10.1016/j.jmpt.2007.04.008. PMID 17574951
- [Background] Moseley GL. Impaired trunk muscle function in sub-acute neck pain: etiologic in the subsequent development of low back pain? Man Ther. 2004 Aug;9(3):157-63. doi: 10.1016/j.math.2004.03.002. PMID 15245710
- [Background] Santana JC. The Serape Effect: A Kinesiological Model for Core Training. Strength & Conditioning Journal. 2003;25(2).
- [Background] Sahrmann S. Movement system impairment syndromes of the extremities, cervical and thoracic spines-e-book: Elsevier Health Sciences; 2010.
- [Background] Kristjansson E, Treleaven J. Sensorimotor function and dizziness in neck pain: implications for assessment and management. J Orthop Sports Phys Ther. 2009 May;39(5):364-77. doi: 10.2519/jospt.2009.2834. PMID 19411769
- [Background] Treleaven J. Sensorimotor disturbances in neck disorders affecting postural stability, head and eye movement control. Man Ther. 2008 Feb;13(1):2-11. doi: 10.1016/j.math.2007.06.003. Epub 2007 Aug 16. PMID 17702636
- [Result] Edmondston S, Bjornsdottir G, Palsson T, Solgard H, Ussing K, Allison G. Endurance and fatigue characteristics of the neck flexor and extensor muscles during isometric tests in patients with postural neck pain. Man Ther. 2011 Aug;16(4):332-8. doi: 10.1016/j.math.2010.12.005. Epub 2011 Jan 20. PMID 21256071
- [Result] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Result] Woby SR, Roach NK, Urmston M, Watson PJ. Psychometric properties of the TSK-11: a shortened version of the Tampa Scale for Kinesiophobia. Pain. 2005 Sep;117(1-2):137-44. doi: 10.1016/j.pain.2005.05.029. PMID 16055269
- [Result] Manske R, Reiman M. Functional performance testing for power and return to sports. Sports Health. 2013 May;5(3):244-50. doi: 10.1177/1941738113479925. PMID 24427396
- [Derived] Dere T, Alemdaroglu-Gurbuz I. Muscular endurance and its association with neck pain, disability, neck awareness, and kinesiophobia in patients with chronic neck pain. Somatosens Mot Res. 2024 Sep;41(3):134-141. doi: 10.1080/08990220.2023.2186390. Epub 2023 Mar 10. PMID 36897182

DOCUMENTS (1):
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/67/NCT05121467/Prot_000.pdf